CLINICAL TRIAL: NCT00789711
Title: A Multicentre, Open-label, Nonrandomised, Non-interventional, Observational Study to Compare Safety and Effectiveness of Biphasic Insulin Aspart 30 (NovoMix 30) and Insulin Detemir (Levemir) for the Treatment of Diabetes Mellitus
Brief Title: An Observational Study to Compare the Safety and Effectiveness of NovoMix® 30 and Levemir™ for the Treatment of Diabetes
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3682
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: biphasic insulin aspart 30
- B
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Evaluation of the safety profile and effectiveness of biphasic insulin aspart 30 in the treatment of diabetes mellitus under normal clinical practice conditions in the Philippines
  Other Names: NovoMix® 30; BIASP
  Groups: A
Drug: insulin detemir — Evaluation of the safety profile and effectiveness of insulin detemir in the treatment of diabetes mellitus under normal clinical practice conditions in the Philippines
  Groups: B

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to compare the clinical safety profile and effectiveness of NovoMix® 30 and Levemir™ for the treatment of diabetes in the Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 1 or type 2 diabetes mellitus
* Patients uncontrolled on oral antidiabetic drugs
* Insulin naïve patients or patients currently on human insulin

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol requirements
* Subjects who are previously enrolled in NovoMix® 30 and Levemir™ study
* Subjects on NovoMix® 30 and Levemir™ therapy
* Subjects with hypersensitivity to NovoMix® 30 or to any of the excipients
* Subjects with hypersensitivity to Levemir™ or to any of the excipients
* Females of child bearing potential who are pregnant, breast feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures are required by local law or practice
* Contraindications and warnings specified in the current prescribing information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with diabetes mellitus who needs insulin treatment at the time of inclusion is eligible for the study, including newly diagnosed subjects who have never received insulin or an insulin analogue before
Sampling Method: Non-Probability Sample
Enrollment: 3131 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of all (Major/Minor/Nocturnal) hypoglycaemic events, reported as serious adverse drug reactions. | during 12 months of treatment

SECONDARY OUTCOMES:
HbA1c | at the end of the study
FBG (Fasting Blood Glucose) | at the end of the study
Average (mean) fasting plasma glucose level | at the end of the study
Number of minor (including nocturnal) hypoglycaemic events | during 12 months of treatment
Number of major (including nocturnal) hypoglycaemic events | during 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manila, Philippines

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com